CLINICAL TRIAL: NCT05948189
Title: Investigation of the Effect of Low Back Health Education on Physical Function and Body Awareness in Academicians: Randomized Controlled Study
Brief Title: Low Back Health Education on Physical Function and Body Awareness in Academicians
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Ugur Cavlak, Clinical Professor, Biruni University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2022/73-06
Record Dates: First submitted 2023-06-16; First posted 2023-07-17 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Low Back Pain, Mechanical
Keywords: Academician; physical function; body awareness; low back health; back school
MeSH Terms: conditions — Low Back Pain | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: 94 (49 female and 45 male) volunteer academicians divided into two groups:intervention group (n=47) and control group (n=47), randomly.
Who Masked: Participant
Masking Description: none of the participants did not know the group they are in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Active Comparator): a 6-week exercise program
  Interventions: Other: exercise program
- Controls (No Intervention): a brochure to read

INTERVENTIONS:
Other: exercise program — The participants of the intervention group received back health education (Back School) in the classroom. After the education program, they participated in exercise training for six weeks (one day a week).
  Arms: intervention group

SUMMARY:
This study was planned to investigate the effect of back health education given to academicians on physical function and body awareness. The participants of the intervention group received back health education (Back School) in the classroom. After the education program, they participated in exercise training for six weeks (one day a week). The control group was only given an informative brochure on back health and asked to read it.

DETAILED DESCRIPTION:
This study was planned to investigate the effect of back health education given to academicians on physical function and body awareness. The study was completed with a total of 94 (49 female and 45 male) volunteer academicians (intervention group n=47, control group n=47) between the ages of 25-65, with a mean age of 43.22±10.924 years. The participants of both groups were evaluated before and after the 6-week education and training. In order to evaluate physical functions of the participants, One Leg Standing Test (eyes open and closed), Half Squat Test, Curl-Up Test, and Sit and Reach Test were used. The Body Awareness Questionnaire (BAQ) was used to assess body awareness of the sample. The participants of the intervention group received back health education (Back School) in the classroom. After the education program, they participated in exercise training for six weeks (one day a week). The control group was only given an informative brochure on back health and asked to read it.

ELIGIBILITY:
Inclusion Criteria:

* Taking part in full-time academic staff at Ondokuz Mayıs University and Samsun University in Turkey.
* To continue his/her career at the university for at least 3 years without break
* Male and female volunteer academicians between the ages of 25-65

Exclusion Criteria:

* Those with any identified back pain problem
* Those who have undergone spinal surgery
* Those with neurological problems
* Those with orthopedic problems
* Those with cardiac or pulmonary problems (except controlled taking by medicines.
* Part-time employees

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2023-06-15 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-10-15 (Actual)

PRIMARY OUTCOMES:
One Leg Standing Test (eyes open and closed) | through study completion, an average of 1 year
  One Leg Standing Test (eyes open and closed)
Half Squat Test | through study completion, an average of 1 year
  performed half squats
Curl-Up Test | through study completion, an average of 1 year
  performed curl-up
Sit and Reach Test | through study completion, an average of 1 year
  participants asked to reach forward on the test table in long sitting position on the mat.
Body Awareness Questionnaire (BAQ) | through study completion, an average of 1 year
  all the participants filled out the questionaire

CONTACTS AND LOCATIONS:
Overall Officials: UGUR CAVLAK, Prof., Principal Investigator — Biruni University
Locations (1):
- Faculty of Health Sciences in Biruni University, Istanbul, Zeytinburnu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: September 1, 2023
Access Criteria: free- open access

REFERENCES:
- [Result] Banerjee S, Argaez C. Multidisciplinary Treatment Programs for Patients with Acute or Subacute Pain: A Review of Clinical Effectiveness, Cost-Effectiveness, and Guidelines [Internet]. Ottawa (ON): Canadian Agency for Drugs and Technologies in Health; 2019 May 7. Available from http://www.ncbi.nlm.nih.gov/books/NBK546002/ PMID 31498579
- [Result] Cortell-Tormo JM, Sanchez PT, Chulvi-Medrano I, Tortosa-Martinez J, Manchado-Lopez C, Llana-Belloch S, Perez-Soriano P. Effects of functional resistance training on fitness and quality of life in females with chronic nonspecific low-back pain. J Back Musculoskelet Rehabil. 2018 Feb 6;31(1):95-105. doi: 10.3233/BMR-169684. PMID 28826168
- [Result] Park HK, Song MK, Kim DJ, Choi IS, Han JY. Comparison of core muscle strengthening exercise and stretching exercise in middle-aged women with fibromyalgia: A randomized, single-blind, controlled study. Medicine (Baltimore). 2021 Dec 17;100(50):e27854. doi: 10.1097/MD.0000000000027854. PMID 34918634